CLINICAL TRIAL: NCT04012853
Title: Remotely Supervised Transcranial Direct Current Stimulation for Persistent Post-traumatic Headache: A Pilot Study
Brief Title: Remotely Supervised tDCS for Persistent Post-traumatic Headache
Acronym: tDCS for PTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3194-P
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-02

CONDITIONS: Persistent Post Traumatic Headache; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- treatment arm (Experimental): tDCS treatment group
  Interventions: Device: transcranial direct current stimulation
- control arm (No Intervention): Sham tDCS

INTERVENTIONS:
Device: transcranial direct current stimulation — Treatment group will receive 20 minutes of tDCS stimulation at 2.0 mA administered daily for five days per week and a total of 4 weeks. During the 20minute treatment session, both treatment and sham groups will complete mindfulness meditation via VA health system approved program (Mindfulness Coach).
  Other Names: tDCS
  Arms: treatment arm

SUMMARY:
This pilot study is designed to provide preliminary data for a large scale, randomized clinical trial to evaluate the efficacy of remotely administrated at home transcranial Direct Current Stimulation (tDCS) with real-time monitoring via VA Tele-health for persistent post traumatic headache associated with mild traumatic brain injury (mTBI). Participants will receive total of 20 sessions of tDCS over four weeks. The investigators anticipate that the results generated from the study will directly translate into immediate meaningful clinical application: not only in management of chronic post traumatic headache, but also in reduction of acute pain medication use, and improving quality of life for our veterans with this debilitating neurological disorder.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the feasibility and efficacy of transcranial Direct Current Stimulation (tDCS) administered at home with real-time monitoring via VA Tele-health for persistent post traumatic headache (PTH) associated with mTBI, and the impact of this treatment on persistent PTH associated functional recovery. Total of 20 participants (10 treatment group, 10 sham control) will be included in this study. The investigators will also evaluate recruitment strategies and participants clinical characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Verified history of mTBI
2. Persistent PTH as defined by International Classification of Headache Disorders (ICHD) III diagnostic criteria("Headache Classification Committee of the International Headache Society (IHS) The ICHD, 3rd Edition 2018).
3. Verification of headache frequency through prospectively collected baseline information during the 28-day screening/baseline phase.
4. Not currently taking a migraine or headache preventive medication OR has been taking a stable dose of a preventive for at least 60 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period.
5. The investigators will include medication overuse headache as defined by ICHD III diagnostic criteria.
6. Participants is either not of childbearing potential, or if they are of childbearing potential, they agree either to remain abstinent or use (or have their partner use) an acceptable method of birth control for the duration of the study.
7. Male or female, age between 20-60 who demonstrates compliance with the electronic Daily Headache Diary during the 28-day baseline phase as defined by entry of headache data on a minimum of 22 to 28 days (80% diary compliance).

Exclusion Criteria:

1. Unable to complete headache diary as required by protocol.
2. Any psychiatric condition with psychotic features, and/or any other psychiatric disorder not stable or well controlled, that would interfere in the ability to complete study activities
3. Received onabotulinumtoxinA, cognitive behavior therapy, physical therapy or any other form of non-pharmacological therapy for headaches during the 4 months before screening.
4. Has a planned military deployment within the 6 months post screening.
5. Active substance abuse within last 4 months.
6. History of seizure, stroke, multiple sclerosis or other unstable neurological condition or a significant abnormal neurological examination.
7. Unable to tolerate tDCS stimulation.
8. Have any other conditions that in the judgment of the Investigator would make the participants unsuitable for inclusion or interfere with participating or completing the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao M. Androulakis, MD, Principal Investigator — Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC
Locations (1):
- Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charvet L, Harrison AT, Mangold K, Moore RD, Guo S, Zhang J, Datta A, Androulakis XM. Remotely supervised at-home tDCS for veterans with persistent post-traumatic headache: a double-blind, sham-controlled randomized pilot clinical trial. Front Neurol. 2023 May 5;14:1184056. doi: 10.3389/fneur.2023.1184056. eCollection 2023. PMID 37213913

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed a 28-day baseline period in which they completed daily headache diaries to validate diagnosis of PPTH.
Groups:
- Treatment Arm: Active tDCS group
  The active tDCS treatment group will receive 20 minutes of tDCS stimulation at 2.0 mA administered daily for five days per week and a total of 4 weeks. During the 20 minute treatment session, they will also complete mindfulness meditation via VA health system approved program (Mindfulness Coach).
- Control Arm: Sham tDCS group
  Sham group will receive 20 minutes of sham tDCS stimulation administered daily for five days per week and a total of 4 weeks. During the 20 minute treatment session, they will also complete mindfulness meditation via VA health system approved program (Mindfulness Coach).
Period: Overall Study
Arm/Group | Treatment Arm | Control Arm
Started | 13 | 13
Completed | 10 | 12
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Unable to tolerate target tDCS intensity | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants were randomly assigned to either the Treatment arm or the Control arm after successful completion of a 28-day baseline period. During this periods participants completed daily headache diaries to establish baseline headache characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (9.2) | 42.2 (8.4) | 45.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 11 | 11 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 8 | 13
  Black of African American | 8 | 5 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 26
Marital Status [Count of Participants; unit: Participants]
  Married | 9 | 9 | 18
  Divorce | 3 | 2 | 5
  Never Married/Domestic Partnership | 1 | 2 | 3
Education Level [Count of Participants; unit: Participants]
  High School Graduate or GED | 2 | 1 | 3
  Some College or Technical School | 4 | 8 | 12
  Bachelor's Degree or Higher | 7 | 4 | 11
Employment Status [Count of Participants; unit: Participants]
  Employed (Full or Part-Time) | 5 | 8 | 13
  Unemployed | 3 | 1 | 4
  Disabled | 2 | 2 | 4
  Retired | 3 | 2 | 5
Number of Headache Days (out of 28 days) [Mean (Standard Deviation); unit: days] | 25.2 (3.7) | 23.8 (4.8) | 24.5 (4.2)
Number of Moderate-to-Severe Headache Days (out of 28 days) [Mean (Standard Deviation); unit: days] | 16.9 (8.3) | 14.8 (6.4) | 16.0 (7.4)
Days of Acute Pain Medication Use (out of 28 days) [Mean (Standard Deviation); unit: days] | 11.5 (11.3) | 9.6 (7.9) | 10.5 (9.4)
Medication overuse [Count of Participants; unit: Participants] | 4 | 4 | 8
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — scale range from 0 to 27, with higher scores indicating more severe depression symptoms
  units on a scale | 14.3 (6.8) | 14.3 (4.6) | 14.3 (5.5)
Headache Impact Test (HIT-6) [Mean (Standard Deviation); unit: units on a scale] — scale range from 36 to 78, with higher scores indicating more substantial functional impairment
  units on a scale | 64.2 (6.4) | 63.2 (7.7) | 63.6 (7.0)
Beck's Anxiety Inventory (BAI) [Mean (Standard Deviation); unit: units on a scale] — scale range from 0 to 63, with higher score indicating greater anxiety
  units on a scale | 31.6 (16.2) | 22.1 (10.1) | 26.4 (13.8)
DSM-5 PTSD Checklist (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — scale range from 0 to 80, with a lower score suggesting a lower incidence of PTSD
  units on a scale | 46.2 (20.0) | 42.7 (19.2) | 44.3 (19.2)
Insomnia Sleep Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — scale range from 0 to 28, with higher scores indicating increased severity of insomnia
  units on a scale | 17.8 (8.5) | 17.7 (6.7) | 17.7 (7.4)
Rivermead Post-Concussion Questionnaire (RPQ) [Mean (Standard Deviation); unit: units on a scale] — scale range from 0 to 64, with higher scores indicating a worse outcome
  units on a scale | 42.0 (13.0) | 42.0 (10.0) | 42.0 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Moderate-to-Severe Headache Days Per Month
Description: To evaluate the improvement in numbers of moderate to severe headache days per month from baseline period to end of treatment phase, and to the end of follow-up phase
Time Frame: Baseline (four-week daily headache diary), following four-week treatment phase, and four week post-treatment follow-up (12 weeks total)
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Mean (Standard Deviation); unit: Days per Month
Groups:
- Control Arm: Sham tDCS group
  Sham group will receive 20 minutes of sham tDCS stimulation administered daily for five days per week and a total of 4 weeks. During the 20 minute treatment session, they will also complete mindfulness meditation via VA health system approved program (Mindfulness Coach).
  * 1 participant was excluded due to being an outlier on multiple measures
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
Days per Month
  End of Treatment (change from baseline) | -2.5 (3.5) | 2.3 (3.5)
  End of Follow-up (change from baseline) | -3.9 (6.5) | 1.2 (6.5)

2. Secondary Outcome: Change From Baseline in the Total Number of Headache Days Per Month
Description: To evaluate improvement in total number of headache days per month, acute pain mediation used based on number of doses of medication taken from baseline period to end of treatment phase, and to end of follow-up phase in the same cohort.
Time Frame: as for outcome 1
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
days per month
  End of Treatment (change from baseline) | -4.0 (5.2) | 1.54 (3.8)
  End of Follow-up (change from baseline) | 2.1 (7.2) | -0.2 (4.4)

3. Secondary Outcome: Change From Baseline in the Quality of Life Based on Change in Headache Impact Test-6 (HIT-6)
Description: To evaluate the impact of headaches on the quality of life measures (pain and disability) based on change in Headache impact test-6 (HIT-6) from baseline period to end of treatment phase, and to end of follow-up phase in persistent PTH. The six-item Headache Impact Test (HIT-6) provides a global measure of adverse headache impact and was developed to use in screening and monitoring patients with headaches in both clinical practice and clinical research. A total HIT-6 score ranges from 36 to 78: Little or no impact = HIT-6 score 49 or less; Some impact = HIT-6 score 50-55; Substantial impact = HIT-6 score 56-59; Severe impact = HIT-6 score 60.
Time Frame: as for outcome 1
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
units on a scale
  End of Treatment (change from baseline) | -4.5 (6.5) | -4.0 (7.3)
  End of Follow-up (change from baseline) | 0.8 (5.4) | -5.4 (18.4)

4. Secondary Outcome: Change From Baseline in the Acute Pain Medication Days Per Month
Description: change in days of acute pain medication use based on number of days taken during the baseline period to end of the treatment and follow up phase
Time Frame: Change from baseline (four-week daily headache diary) following four-week treatment phase and four week post-treatment follow-up (12 weeks total)
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Mean (Standard Deviation); unit: Days of Medication Use per Month
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
Days of Medication Use per Month
  End of Treatment (change from baseline) | -2.7 (4.2) | -0.4 (3.7)
  End of Follow-up (change from baseline) | 3.0 (6.4) | -2.3 (10.2)

5. Secondary Outcome: Number of Participants With a 50% Reduction in Headache Frequency
Description: Number of participants with 50% or more reduction in monthly headache days (compared to baseline) will be evaluated.
Time Frame: as for outcome 1
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
Participants
  End of Treatment: 50% or greater reduction in headache days | 1 | 0
  End of Treatment: Less than 50% reduction in headache days | 9 | 11
  End of Follow-up: 50% or greater reduction in headache days | 2 | 0
  End of Follow-up: Less than 50% reduction in headache days | 8 | 11

6. Secondary Outcome: Change From Baseline in Scores on the Patient Health Questionnaire (PHQ-9)
Description: assess changes in patient reported depression severity - scale range from 0 to 27, with higher scores indicating more severe depression symptoms
Time Frame: as for outcome 1
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
score on a scale
  End of Treatment (change from baseline) | -0.6 (4.1) | 0.1 (4.4)
  End of Follow-up (change from baseline) | 0.1 (4.2) | -1.0 (5.6)

7. Secondary Outcome: Change From Baseline in Scores on the DSM-5 PTSD Checklist (PCL-5)
Description: Assess changes in patient reported PTSD-like symptoms - scale range from 0 to 80, with a lower score suggesting a lower incidence of PTSD
Time Frame: as for outcome 1
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
score on a scale
  End of Treatment (change from baseline) | 2.9 (9.3) | 1.9 (7.4)
  End of Follow-up (change from baseline) | -1.4 (17.2) | -1.5 (12.4)

8. Secondary Outcome: Change From Baseline in Scores on the Beck's Anxiety Inventory (BAI)
Description: Assess changes in patient reported anxiety - scale range from 0 to 63, with higher score indicating greater anxiety
Time Frame: as for outcome 1
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
score on a scale
  End of Treatment (change from baseline) | -3.2 (8.6) | 1.9 (10.5)
  End of Follow-up (change from baseline) | -2.8 (9.6) | 3.5 (10.8)

9. Secondary Outcome: Change From Baseline in Scores on the Rivermead Post-Concussion Questionnaire (RPQ)
Description: Assess changes in patient reported concussion-related symptoms - scale range from 0 to 64, with higher scores indicating a worse outcome
Time Frame: Change from baseline following four-week treatment phase and four week post-treatment follow-up (8 weeks total)
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
score on a scale
  End of Treatment (change from baseline) | -10.2 (19.1) | -4.2 (11.7)
  End of Follow-up (change from baseline) | -4.8 (10.6) | -4.0 (14.8)

10. Secondary Outcome: Change From Baseline in Scores on the Insomnia Severity Index (ISI)
Description: Assess changes in patient reported insomnia/sleep disturbances - scale range from 0 to 28, with higher scores indicating increased severity of insomnia
Time Frame: as for outcome 1
Population: Analysis was conducted on participants completing post-treatment, and follow-up evaluations
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 10 | 11
score on a scale
  End of Treatment (change from baseline) | -0.5 (5.5) | 0.2 (5.1)
  End of Follow-up (change from baseline) | -0.5 (4.2) | 0.9 (8.4)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded following each daily session over the course of the four-week treatment phase (20-sessions).
Description: Following each treatment session, in clinic or at-home, the supervisor would ask each participant to report whether they experienced (yes/no) any side-effects from a standardized list.
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 8/10 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=10) | Control Arm (N=12)
Tingling Sensation (Skin and subcutaneous tissue disorders) | 7 | 11 — Tingling sensation beneath tDCS electrode
Prickling Sensation (Skin and subcutaneous tissue disorders) | 1 | 2 — Prickling sensation beneath tDCS electrode
Warming Sensation (Skin and subcutaneous tissue disorders) | 3 | 7 — Warming sensation beneath the tDCS electrode
Itching (Skin and subcutaneous tissue disorders) | 2 | 3 — Itching beneath the tDCS electrode
Redness/Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 0 — Redness or dry skin beneath the tDCS electrode
Numbing Sensation (Skin and subcutaneous tissue disorders) | 1 | 1 — Numbness beneath the tDCS electrode
Pulsing/Throbbing (General disorders) | 1 | 1 — Pulsing of throbbing sensation beneath the tDCS electrode
Dizziness/Lightheaded (General disorders) | 1 | 1 — Feeling dizzy or lightheaded during/after treatment session
Vertigo (General disorders) | 0 | 1 — Feeling of vertigo during/after treatment session
Fatigue (General disorders) | 0 | 1 — Feeling of increased fatigue during/after treatment session
Other (General disorders) | 2 | 4 — Feeling one of the following during/after treatment: pain, sharp sensations, back pain, pressure, and/or eye twitches (each reported by <= 1 participant)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT04012853/Prot_001.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT04012853/SAP_002.pdf
  • Informed Consent Form (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT04012853/ICF_000.pdf